CLINICAL TRIAL: NCT00564395
Title: Role of Insulin Aspart and Detemir to Assess Glucose Excursion in Children With Type 1 Diabetes
Brief Title: Detemir: Role in Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Rubina Heptulla, Principal Investigator, Montefiore Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-16541
Record Dates: First submitted 2007-11-27; First posted 2007-11-28 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: blood sugar; glycemic
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin Detemir+RAI, then Insulin Detemir and RAI separately (Experimental): Participants first received, Insulin Detemir mixed with RAI, twice daily as subcutaneous injection for 10 days. Then they received Insulin Detemir and RAI as separate subcutaneous injections, twice daily for the next 10 days.
  Interventions: Drug: Insulin Detemir mixed with RAI injection
- Insulin Detemir and RAI separately, then Insulin Detemir+RAI (Active Comparator): Participants first received Insulin Detemir and RAI as separate subcutaneous injections, twice daily for 10 days. Then they received Insulin Detemir mixed with RAI, twice daily as subcutaneous injection for the next 10 days.
  Interventions: Drug: Insulin Detemir and RAI injection

INTERVENTIONS:
Drug: Insulin Detemir mixed with RAI injection — Insulin Detemir mixed with RAI injection is given twice daily as subcutaneous injection
  Arms: Insulin Detemir+RAI, then Insulin Detemir and RAI separately
Drug: Insulin Detemir and RAI injection — Insulin detemir and RAI are given as separate injections, twice daily as subcutaneous injection
  Arms: Insulin Detemir and RAI separately, then Insulin Detemir+RAI

SUMMARY:
Study of blood sugars in the children with Type 1 Diabetes Mellitus (T1DM), who are given insulin detemir and a rapid acting insulin (aspart). It is hypothesized that there is no difference in the patterns of blood sugars when detemir is given in the same syringe or in separate syringes with rapid acting insulin.

DETAILED DESCRIPTION:
One of the barriers to good glycemic control in children with type 1 diabetes is multiple daily insulin injections. Mixing rapid-acting (detemir) and slow- acting insulins (aspart) in the same syringe would decrease the number of injections and may improve adherence

This study hypothesized that slow-acting insulin detemir mixed with aspart would have equivalent effects on blood glucose versus giving them as separate injections in children with type 1 diabetes.

Eighteen pediatric subjects with type 1 diabetes (11 males and 7 females) were recruited. However only 14 subjects completed this 20-day, randomized, crossover, and open-labeled study. The subjects were randomly assigned to either Study A (both insulin detemir and rapid acting insulin (RAI)) or Study B (either detemir or aspart) for the first 10 days. They were then crossed over for the last 10 days. Each subject underwent 72 h of continuous glucose monitoring (CGM) during the last 72 h, for both Study A and Study B.Data of 48 h from midnight of the 1st day to mid- night of the 3rd day of the 72-h (CGM) were used for analysis to ensure the same starting and ending times of monitoring for all subjects.Sustained glucose values over time were calculated as area under the curve (AUC), index of blood glucose control as M-value and glucose excursion as mean amplitude of glucose excursion (MAGE)

ELIGIBILITY:
Inclusion Criteria:

* Subjects with antibody positive Type 1 Diabetes Mellitus (T1DM)
* On insulin glargine for at least 3 months
* Age 10-25 years
* Not on medications that may affect glucose concentrations
* Hemoglobin A1C (HbA1C) of less than 9 %
* Body Mass Index (BMI) less than 95th % and more than 10th%
* Supportive family

Exclusion Criteria:

* Subjects with undetermined diabetes or Type 2 Diabetes Mellitus (T2DM)
* Unable to adhere to insulin regimen
* Positive urine pregnancy test

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2007-08; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rubina A Heptulla, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital Endocrine and Diabetes Clinic, Houston, Texas, United States

REFERENCES:
- [Background] Nguyen TM, Renukuntla VS, Heptulla RA. Mixing insulin aspart with detemir does not affect glucose excursion in children with type 1 diabetes. Diabetes Care. 2010 Aug;33(8):1750-2. doi: 10.2337/dc10-0169. Epub 2010 May 26. PMID 20504899

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighteen participants were recruited for this trial. However, only 14 participants completed both study visits. Subjects were recruited from the clinics through fliers and online postings
Pre-assignment Details: One male subject dropped out because of a very active sports schedule and could not continue participation.
  Three subjects (two males and one female) had trouble with the Continuous Glucose Monitoring (CGM) tracing and, therefore, were excluded from the final analysis.
Period: First Intervention (10 Days)
Arm/Group | Insulin Detemir+RAI, Then Insulin Detemir and RAI Separately | Insulin Detemir and RAI Separately, Then Insulin Detemir+RAI
Started | 9 | 9
Received Intervention | 7 | 7
Completed | 7 | 7
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Trouble with the CGM tracing | 1 | 2
Period: Second Intervention (10 Days)
Arm/Group | Insulin Detemir+RAI, Then Insulin Detemir and RAI Separately | Insulin Detemir and RAI Separately, Then Insulin Detemir+RAI
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to receive either Insulin Detemir mixed with RAI subcutaneous injection twice daily or Insulin Detemir and RAI as separate subcutaneous injections, twice daily
Arm/Group | All Study Participants
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.8 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Assess the Mean Area Under the Curve (AUC) for Blood Glucose Concentration in Subjects Treated With Either Insulin Detemir Mixed With Rapid Acting Insulin (RAI) or Insulin Detemir and RAI as Separate Subcutaneous Injections
Description: Blood glucose concentration in terms of mean AUC (0-48 hours)was determined in subjects treated with either Insulin Detemir mixed with RAI or Insulin Detemir and RAI as separate subcutaneous injections.
Time Frame: 0-48 hours post-dose
Measure: Mean (Standard Deviation); unit: mmol*hr/L
Groups:
- Insulin Detemir Mixed With RAI Injection: Participants who received Insulin Detemir mixed with RAI injection, twice daily as subcutaneous injection in either the first or last 10 days of the study.
- Insulin Detemir and RAI Injection Separately: Participants who received Insulin Detemir and RAI as separate subcutaneous injections, twice daily in either the first or last 10 days of the study.
Arm/Group | Insulin Detemir Mixed With RAI Injection | Insulin Detemir and RAI Injection Separately
Number analyzed (Participants) | 14 | 14
mmol*hr/L | 457 (70) | 469 (112)

ADVERSE EVENTS:
Time Frame: 10 days for each intervention
Groups:
- Insulin Detemir Mixed With RAI Injection: Participants who received Insulin Detemir mixed with RAI, twice daily as subcutaneous injection for 10 days.
- Insulin Detemir and RAI Injection Separately: Participants who received Insulin Detemir and RAI as separate subcutaneous injections, twice daily for 10 days.
Arm/Group | Insulin Detemir Mixed With RAI Injection | Insulin Detemir and RAI Injection Separately
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No